CLINICAL TRIAL: NCT02497183
Title: Impact of Presence of Oral Contrast Material in the Large Intestine on the Recognition of Appendix During an Ultrasound Exam
Brief Title: Impact of Oral Contrast in the Large Intestine on the Recognition of Appendix
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0053-15-EMC
Record Dates: First submitted 2015-06-25; First posted 2015-07-14 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- first (Experimental): a repeat abdominal ultrasound exam to patients following the filling of bowel with contrast material per os.
  Interventions: Device: ultrasound; Other: iodine based solution of oral contrast material

INTERVENTIONS:
Device: ultrasound — A repeat ultrasound exam following oral contrast material consumption
Other: iodine based solution of oral contrast material — A solution of oral contrast material that is routinely used in our institution prior to performing a computed tomographic (CT) examinations of the gastrointestinal tract will be given prior to performing the repeat ultrasound/
  Other Names: Telebrix Gastro

SUMMARY:
Acute appendicitis is the most common cause of abdominal pain requiring surgical intervention.

The gold standard test for the diagnosis of acute appendicitis is the CT scan. Despite its effectiveness, the test involves exposure to a high dose of radiation.

Using ultrasound to diagnose this condition has been described extensively in the medical literature, and this test has a very high specificity (over 95%), however sensitivity of the test is not as good and varies between 40% and 90%. Major limitations of the Ultrasound test include operator dependency as well as factors such as body habitus of the patient, presence of technical disturbances (artifacts) caused by gas in the large intestine and inadequate cooperation from the patient during the exam. All of these factors may affect the ability to detect sonographic signs of appendicitis.

The investigators believe that it is possible to reduce the amount of artifacts caused by the presence of gas in the intestine by filling of the colon with liquid suspension that is routinely given in the investigators' hospital before performing an abdominal CT and performing an additional ultrasound scan to those patients in which the initial ultrasound examination (without any preparation) proved to be equivocal or not diagnostic.

The target population for the study is any patient who arrives to the emergency room with complaints of right lower quadrant abdominal pain and it is decided by the referring physician in the ER to start diagnostic workup for suspected appendicitis by performing an ultrasound, if the ultrasound exam proves to be equivocal or not diagnostic and it is decided that the patient needs to continue investigation by performing a CT scan, the patient will receive contrast material orally for approximately 180 minutes and prior to the CT the investigators intend to repeat the ultrasound. The investigators hypothesize that the repeat ultrasound will allow a statistically significant improvement in the detection rate of the appendix.

DETAILED DESCRIPTION:
Acute appendicitis is the most common cause of abdominal pain requiring surgical intervention.

The gold standard test for the diagnosis of acute appendicitis is the CT scan. Despite its effectiveness, the test involves exposure to a high dose of radiation.

Using ultrasound to diagnose this condition has been described extensively in the medical literature, and this test has a very high specificity (over 95%), however sensitivity of the test is not as good and varies between 40% and 90%. Major limitations of the Ultrasound test include operator dependency as well as factors such as body habitus of the patient, presence of technical disturbances (artifacts) caused by gas in the large intestine and inadequate cooperation from the patient during the exam. All of these factors may affect the ability to detect sonographic signs of appendicitis.

The investigators believe that it is possible to reduce the amount of artifacts caused by the presence of gas in the intestine by filling of the colon with liquid suspension that is routinely given in the investigators' hospital before performing an abdominal CT and performing an additional ultrasound scan to those patients in which the initial ultrasound examination (without any preparation) proved to be equivocal or not diagnostic.

The target population for the study is any patient who arrives to the emergency room with complaints of right lower quadrant abdominal pain and it is decided by the referring physician in the ER to start diagnostic workup for suspected appendicitis by performing an ultrasound, if the ultrasound exam proves to be equivocal or not diagnostic and it is decided that the patient needs to continue investigation by performing a CT scan, the patient will receive contrast material orally for approximately 180 minutes and prior to the CT the investigators intend to repeat the ultrasound. The investigators hypothesize that the repeat ultrasound will allow a statistically significant improvement in the detection rate of the appendix.

expected number of recruited patients: 200

ELIGIBILITY:
Inclusion Criteria:

* age 14 years to 120 years
* patients that underwent an ultrasound exam that proved to be equivocal or not diagnostic
* patients who were sent to perform a CT scan that includes drinking oral contrast material.

Exclusion Criteria:

* pregnant patients
* patients with known allergy to oral contrast material (TELEBRIX gastro)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
statistically significant improvement in the detection rate of the appendix | one year
  ultrasound exam with filling of the colon with liquid suspension will allow a statistically significant improvement in the detection rate of the appendix compared to an exam without any preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Roshkovan, M.D, Study Chair — haemek medical center
Locations (1):
- HaEmek medical center, Afula, Israel